CLINICAL TRIAL: NCT06376175
Title: Task Atlas: An Observational Study to Develop a Task Atlas of Brain Recruitment During a Digital Game-based Program
Brief Title: Task Atlas: Study to Develop a Task Atlas of Brain Recruitment During a Digital Game-based Program
Status: Completed | Type: Observational
Sponsor: Lumos Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LL-016
Record Dates: First submitted 2024-04-03; First posted 2024-04-19 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Healthy Adults
Keywords: cognition; fMRI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthy volunteers ages 25-40 from the general US population who meet the eligibility criteria and are enrolled will (a) play Lumosity games at least 20 times each in under 60 days and (b) then complete one session of task-based functional magnetic resonance imaging (fMRI) while playing Lumosity games.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 25-40 years of age.
* Ability to understand and speak English, follow written and verbal instructions (English), and give informed consent (English), as assessed by the PI or project manager.
* Ability to comply with all the testing and study requirements, including the ability to independently complete daily, online Lumosity games on a reliable, internet-connected device.
* Geographical location within 100 miles of the study imaging center.

Exclusion Criteria:

* Current, controlled (requiring treatment) or uncontrolled psychiatric diagnosis, including but not limited to posttraumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder, conduct disorder, attention- deficit/hyperactivity disorder, or other symptomatic manifestations that in the opinion of the PI may confound study data/assessments.
* Current, controlled (requiring treatment) or uncontrolled neurological diagnosis, including but not limited to Alzheimer's Disease, other dementias, mild cognitive impairment, Huntington's Disease, Parkinson's Disease, multiple sclerosis, stroke, epilepsy, aphasia, or other condition that in the opinion of the PI may confound study data/assessments.
* Any other medical condition in the last 90 days that in the opinion of the PI may confound study data/assessments.
* Has been under the care of a caretaker or has not been living independently in the last 90 days.
* In the last three years has used online brain training programs (e.g., BrainHQ, Lumosity, Peak) for more than two weeks continuously.
* Known sensitivity (such as headaches, dizziness, nausea) to bright, stimulating video displays.
* History of seizures (excluding febrile seizures), or significant motor or vocal tics, including but not limited to Tourette's Disorder and photo-sensitive epilepsy.
* Visual acuity that cannot be corrected that prevents or negatively impacts computer activity.
* Pregnancy, or strong likelihood of pregnancy.
* Left-handed or ambidextrous.
* Unwillingness or inability to comply with imaging safety protocols. Inability includes but is not limited to metal implants or exposure to shrapnel.
* Any other condition that in the opinion of the PI may confound study data.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults age 25-40
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
BOLD response during gameplay | Day 60
  Whole-brain blood oxygen level-dependent (BOLD) response during gameplay
Responder rates | Day 60
  Percentage of participants who show A) BOLD response by brain region during gameplay, B) Between-network connectivity, based on BOLD responses, during gameplay, C) Within-network connectivity, based on BOLD responses, during gameplay
Structural MRI volumetrics: Volume | Day 60
  Volume at rest
Structural MRI volumetrics: Cortical thickness | Day 60
  Cortical thickness measured in millimeters
Structural MRI volumetrics: Brain-Predicted Age Difference | Day 60
  Brain-Predicted Age Difference at rest
Behavior response: Game score | Day 60
  Score on game after completion of gameplay
BAMS-7 (Brief Attention and Mood Scale of 7 Items) | Day 60
  Subject-reported BAMS-7 (Brief Attention and Mood Scale of 7 Items) including the Attention subscale, Mood subscale, and Total, measured post-imaging
VGPQ (Video Game Playing Questionnaire) | Day 60
  Subject-reported VGPQ (Video Game Playing Questionnaire) including non-video game playing (NVGP) and video game playing (VGP)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Madore, PhD, Principal Investigator — Lumos Labs, Inc.
Locations (1):
- UC Davis Imaging Research Center (IRC), Sacramento, California, United States